CLINICAL TRIAL: NCT06446505
Title: Feasibility, Acceptability, and Effectiveness of an Online Decision Aid for Patients With Parkinson's Disease Considering Deep Brain Stimulation Surgery Using a Pragmatic, Randomized Pilot Trial
Brief Title: Evaluation of a Decision Aid for Deep Brain Stimulation Surgery for Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-2390; K12AR084226 (NIH)
Record Dates: First submitted 2024-05-22; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; Decision Aid
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Decision Aid (Experimental): Participants will receive the Decision Aid at baseline.
  Interventions: Other: Deep Brain Stimulation Decision Aid
- Delayed Decision Aid (Active Comparator): Participants will receive the Decision Aid at the end of the deep brain stimulation surgery evaluation process.
  Interventions: Other: Deep Brain Stimulation Decision Aid

INTERVENTIONS:
Other: Deep Brain Stimulation Decision Aid — An online decision support tool that provides education about deep brain stimulation and the alternatives, and includes value clarification exercise.

SUMMARY:
The goal of this clinical trial is to learn if a Decision Aid can help patients with Parkinson's disease make a decision about undergoing Deep Brain Stimulation surgery. The main questions it aims to answer are:

* Is the Decision Aid acceptable to patients with Parkinson's disease considering Deep Brain Stimulation surgery?
* Does the decision aid improve decision quality (informed, value-based decision) and uncertainty about the decision?

Researchers will compare immediate use of the decision aid during the evaluation process for deep brain stimulation surgery to delayed introduction of the decision aid.

Participants will:

* Receive the decision aid at the beginning of the evaluation process or towards the end
* Complete surveys at 5 visits (remote or in-person) over approximately 6 months

ELIGIBILITY:
Inclusion Criteria:

* Adults with a diagnosis of Parkinson's disease referred for deep brain stimulation surgery evaluation at the University of Colorado

Exclusion Criteria:

* Atypical Parkinsonism
* Diagnosis of Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Acceptability tool from the Ottawa Hospital Research Institute | Baseline
  This tool measures the comprehensibility of components of the decision aid including its length, amount of information, balance and suitability for decision-making. Higher scores indicate that the tool is more acceptable.
Acceptability tool from the Ottawa Hospital Research Institute | 2 weeks after decision for deep brain stimulation surgery
  This tool measures the comprehensibility of components of the decision aid including its length, amount of information, balance and suitability for decision-making. Higher scores indicate that the tool is more acceptable.
Decisional Conflict Scale (DCS) | Baseline
  The Decisional Conflict Scale measures the perceptions of uncertainty in choosing options, including uncertainty related to feeling uninformed, unclear about personal values and unsupported in decision-making. The minimum score is a 0 and the maximum score is 100. Higher scores indicate more decisional conflict.
Decisional Conflict Scale (DCS) | 1 Month
  The Decisional Conflict Scale measures the perceptions of uncertainty in choosing options, including uncertainty related to feeling uninformed, unclear about personal values and unsupported in decision-making. The minimum score is a 0 and the maximum score is 100. Higher scores indicate more decisional conflict.
Decisional Conflict Scale (DCS) | 3 Months
  The Decisional Conflict Scale measures the perceptions of uncertainty in choosing options, including uncertainty related to feeling uninformed, unclear about personal values and unsupported in decision-making. The minimum score is a 0 and the maximum score is 100. Higher scores indicate more decisional conflict.
Decisional Conflict Scale (DCS) | 2 weeks after decision for deep brain stimulation surgery
  The Decisional Conflict Scale measures the perceptions of uncertainty in choosing options, including uncertainty related to feeling uninformed, unclear about personal values and unsupported in decision-making. The minimum score is a 0 and the maximum score is 100. Higher scores indicate more decisional conflict.
Decisional Conflict Scale (DCS) | 2 months post-Deep brain stimulation surgery or 2 months post decision not to undergo surgery
  The Decisional Conflict Scale measures the perceptions of uncertainty in choosing options, including uncertainty related to feeling uninformed, unclear about personal values and unsupported in decision-making. The minimum score is a 0 and the maximum score is 100. Higher scores indicate more decisional conflict.

SECONDARY OUTCOMES:
Decision Quality Worksheet | 2 weeks after decision for deep brain stimulation surgery
  The worksheet measures how well participants understood the options and outcomes presented in the decision aid, as well as if their decision was consistent with their goals and values. For the knowledge portion of the worksheet, the scores range from 0 to 10, with higher scores indicating increased knowledge about DBS.
Decision Quality Worksheet | 2 months post-Deep brain stimulation surgery or 2 months post decision not to undergo surgery
  The worksheet measures how well participants understood the options and outcomes presented in the decision aid, as well as if their decision was consistent with their goals and values. For the knowledge portion of the worksheet, the scores range from 0 to 10, with higher scores indicating increased knowledge about DBS.
Decision Self-Efficacy scale | Baseline
  This scale measures the participant's self-confidence in or belief in one's ability to make decisions and participate in shared decision-making. The scores range from 0 to 100. A score of 0 means "extremely low self efficacy" and a score of 100 means "extremely high self efficacy".
Decision Self-Efficacy scale | 3 Months
  This scale measures the participant's self-confidence in or belief in one's ability to make decisions and participate in shared decision-making. The scores range from 0 to 100. A score of 0 means "extremely low self efficacy" and a score of 100 means "extremely high self efficacy".
Decision Self-Efficacy scale | 2 weeks after decision for deep brain stimulation surgery
  This scale measures the participant's self-confidence in or belief in one's ability to make decisions and participate in shared decision-making. The scores range from 0 to 100. A score of 0 means "extremely low self efficacy" and a score of 100 means "extremely high self efficacy".
Decision Readiness Instrument | Baseline
  This validated, single-item instrument assesses how ready the participant is to make a decision about deep brain stimulation surgery. The scores vary from 0 "not at all ready" to 5 "completely ready".
Decision Readiness Instrument | 1 Month
  This validated, single-item instrument assesses how ready the participant is to make a decision about deep brain stimulation surgery. The scores vary from 0 "not at all ready" to 5 "completely ready".
Decision Readiness Instrument | 3 Months
  This validated, single-item instrument assesses how ready the participant is to make a decision about deep brain stimulation surgery. The scores vary from 0 "not at all ready" to 5 "completely ready".
Decision Readiness Instrument | 2 weeks after decision for deep brain stimulation surgery
  This validated, single-item instrument assesses how ready the participant is to make a decision about deep brain stimulation surgery. The scores vary from 0 "not at all ready" to 5 "completely ready".
Satisfaction with Decision Scale | 2 weeks after decision for deep brain stimulation surgery
  This scale measures how satisfied the participant is with their decision about whether or not to undergo deep brain stimulation surgery. The areas of satisfaction include how informed they were, if the decision was the best for them, if the decision was consistent with their values and if they had as much input as they wanted. Scores range from 6 to 30. Higher scores indicate higher satisfaction with the decision.
Satisfaction with Decision Scale | 2 months post-Deep brain stimulation surgery or 2 months post decision not to undergo surgery
  This scale measures how satisfied the participant is with their decision about whether or not to undergo deep brain stimulation surgery. The areas of satisfaction include how informed they were, if the decision was the best for them, if the decision was consistent with their values and if they had as much input as they wanted. Scores range from 6 to 30. Higher scores indicate higher satisfaction with the decision.
Parkinson's Disease Quality of Life Questionnaire - 8 (PDQ-8) | Baseline
  This questionnaire measures quality of life in Parkinson's disease related to the 8 dimensions of mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication and bodily discomfort. Scores range from 0 to 100 with higher scores indicating lower quality of life.
Parkinson's Disease Quality of Life Questionnaire - 8 (PDQ-8) | 2 weeks after decision for deep brain stimulation surgery
  This questionnaire measures quality of life in Parkinson's disease related to the 8 dimensions of mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication and bodily discomfort. Scores range from 0 to 100 with higher scores indicating lower quality of life.
Parkinson's Disease Quality of Life Questionnaire - 8 (PDQ-8) | 2 months post-Deep brain stimulation surgery or 2 months post decision not to undergo surgery
  This questionnaire measures quality of life in Parkinson's disease related to the 8 dimensions of mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication and bodily discomfort. Scores range from 0 to 100 with higher scores indicating lower quality of life.
Expectations | Baseline
  Asks participants which Parkinson's symptoms they expect to see improvement in with deep brain stimulation surgery.
Expectations | 1 Month
  Asks participants which Parkinson's symptoms they expect to see improvement in with deep brain stimulation surgery.
Expectations | 3 Months
  Asks participants which Parkinson's symptoms they expect to see improvement in with deep brain stimulation surgery.
Expectations | 2 weeks after decision for deep brain stimulation surgery
  Asks participants which Parkinson's symptoms they expect to see improvement in with deep brain stimulation surgery.
Shared Decision-Making Questionnaire - 9 | 1 Month
  This questionnaire measures the degree of shared decision-making that took place in physician visits discussing deep brain stimulation surgery. The scores range from 0 (no perceived shared decision-making) to 100 (highest level of perceived shared decision-making).
Shared Decision-Making Questionnaire - 9 | 3 Months
  This questionnaire measures the degree of shared decision-making that took place in physician visits discussing deep brain stimulation surgery. The scores range from 0 (no perceived shared decision-making) to 100 (highest level of perceived shared decision-making).
Shared Decision-Making Questionnaire - 9 | 2 weeks after decision for deep brain stimulation surgery
  This questionnaire measures the degree of shared decision-making that took place in physician visits discussing deep brain stimulation surgery. The scores range from 0 (no perceived shared decision-making) to 100 (highest level of perceived shared decision-making).
Trust in the Surgeon Scale | 2 weeks after decision for deep brain stimulation surgery
  This scale measures how much the participant trusts their surgeon. The scale ranges from 11 to 55, with higher scores indicating a higher level of trust.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle E Fullard, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
We plan to share the de-identified dataset after the primary results have been accepted for publication. No patient identifiers will be included in the shared data.